CLINICAL TRIAL: NCT01264744
Title: Concordance Study for Detection of Chromosomal Aberrations Using FISH in Urine Samples Sections
Brief Title: Detection of Chromosomal Aberrations in Urine Samples Using Fluorescent in Situ Hybridization (FISH) (UroVysion Test)
Status: Completed | Type: Observational
Sponsor: Applied Spectral Imaging Ltd. (Industry)
Responsible Party: Nir Katzir, Applied Spectral Imaging Ltd.
Other Study IDs: ASI-UroF
Record Dates: First submitted 2010-12-21; First posted 2010-12-22 (Estimated); Last update posted 2010-12-23 (Estimated); Status verified 2010-12

CONDITIONS: Bladder Cancers
Keywords: Bladder cancer; Chromosomal aberrations; FISH; Urine sample
MeSH Terms: conditions — Urinary Bladder Neoplasms; Chromosome Aberrations

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Urine samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is the identification of chromosomal aberrations in urine samples.

The imaging system is intended for diagnostic use as an aid to the pathologist in the detection, counting and classification of UroVysion FISH stained Urine samples.

DETAILED DESCRIPTION:
The FISH test detect chromosomal aberrations in urine specimens from persons with hematuria suspected of having bladder cancerous using the UroVysion® Bladder Cancer Kit (UroVysion Kit) which is FDA approved. This kit is designed to detect aneuploidy for chromosomes 3, 7, 17, and loss of the 9p21 locus. Results from the UroVysion Kit are intended for use, in conjunction with and not in lieu of current standard diagnostic procedures, as an aid for initial diagnosis of bladder carcinoma in patients with hematuria and subsequent monitoring for tumor recurrence in patients previously diagnosed with bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* Well stained slides with bright FISH signals

Exclusion Criteria:

* Very old slides that were already bleached

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with hematuria that are suspected in having bladder carcinoma, and in patients previously diagnosed with bladder cancer.
Sampling Method: Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2009-11; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheila - Dobin, Ph.D., Study Director — Section Chief, Cytogenetics
Locations (3):
- United States (3):
  - VA Hospital, Los Angeles, California
  - PLUS Diagnostics, Union, New Jersey
  - Sheila Dobin, Ph.D., Temple, Texas